CLINICAL TRIAL: NCT07268430
Title: A Multicenter, Randomized, Open-Label, Parallel-Group, Multiple-Dose Bioequivalence Study of Paliperidone Palmitate Injection in Chinese Patients With Schizophrenia
Brief Title: Bioequivalence Study of Long-Acting Paliperidone Palmitate in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYHF2036-001
Record Dates: First submitted 2025-09-30; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paliperidone Palmitate 1-Month Formulation (PP1M) (Test Group) (Experimental): Participants will receive paliperidone palmitate injection manufactured by CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd., administered intramuscularly. Dosing regimen: 150 mg on Day 1 and 100 mg on Day 8, followed by 100 mg every 28 days (starting Day 1 regimen); or 100 mg every 28 days (starting Day 36 regimen).
  Interventions: Drug: Paliperidone Palmitate Injection(PP1M); Drug: Paliperidone Palmitate Injection(PP1M)(Reference Group)
- Paliperidone Palmitate 1-Month Formulation (PP1M) (Reference Group) (Active Comparator): Participants will receive paliperidone palmitate injection (Invega Sustenna®) manufactured by Janssen Pharmaceutica N.V., administered intramuscularly. Dosing regimen: 150 mg on Day 1 and 100 mg on Day 8, followed by 100 mg every 28 days (starting Day 1 regimen); or 100 mg every 28 days (starting Day 36 regimen).
  Interventions: Drug: Paliperidone Palmitate Injection(PP1M); Drug: Paliperidone Palmitate Injection(PP1M)(Reference Group)

INTERVENTIONS:
Drug: Paliperidone Palmitate Injection(PP1M) — Paliperidone palmitate injection will be administered intramuscularly according to two dosing regimens based on participants' prior exposure to paliperidone palmitate:
  1. Participants with no prior use of paliperidone palmitate injection, or whose last dose was administered more than 6 months ago (for the once-monthly formulation), or more than 5 half-lives ago (for the once-every-3-months formulation):
     Day 1: 150 mg, deltoid muscle Day 8: 100 mg, deltoid muscle Followed by 100 mg every 28 days thereafter Approximate treatment duration: 148 days
  2. Participants who have previously received at least 3 injections (including 150 mg Day 1 loading dose and 100 mg Day 8 loading dose, deltoid muscle) of the once-monthly formulation (100 mg) of paliperidone palmitate and whose last dose was given within 4 to 6 weeks prior to enrollment:
  Continue with 100 mg every 28 days Approximate treatment duration: 113 days
  Other Names: SYHF2036
Drug: Paliperidone Palmitate Injection(PP1M)(Reference Group) — Paliperidone palmitate injection will be administered intramuscularly according to two dosing regimens based on participants' prior exposure to paliperidone palmitate:
  1. Participants with no prior use of paliperidone palmitate injection, or whose last dose was administered more than 6 months ago (for the once-monthly formulation), or more than 5 half-lives ago (for the once-every-3-months formulation):
     Day 1: 150 mg, deltoid muscle Day 8: 100 mg, deltoid muscle Followed by 100 mg every 28 days thereafter Approximate treatment duration: 148 days
  2. Participants who have previously received at least 3 injections (including 150 mg Day 1 loading dose and 100 mg Day 8 loading dose, deltoid muscle) of the once-monthly formulation (100 mg) of paliperidone palmitate and whose last dose was given within 4 to 6 weeks prior to enrollment:
  Continue with 100 mg every 28 days Approximate treatment duration: 113 days
  Other Names: Invega Sustenna

SUMMARY:
This multicenter, randomized, open-label, parallel-group, multiple-dose study is designed to evaluate the bioequivalence, at pharmacokinetic steady state, of a paliperidone palmitate injection manufactured by CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Test Group) and a paliperidone palmitate injection manufactured by Janssen Pharmaceutica N.V. (Reference Group) in patients with schizophrenia in China. Bioequivalence will be assessed based on steady-state pharmacokinetic parameters after repeated intramuscular administration (e.g., Cmax,ss and AUCτ). The safety and tolerability of the test and reference products will also be evaluated.

DETAILED DESCRIPTION:
Purpose: This trial was conducted to evaluate the bioequivalence of a test (T) and a reference (R) formulation of once-monthly paliperidone palmitate (PP1M) in patients with schizophrenia.

Patients and methods: In this randomized, open-label, parallel-group, steady-state bioequivalence study, patients with stabilized schizophrenia were randomized 1:1 to receive T or R formulation. The regimen was 150 mg deltoid on Day 1, then 100 mg deltoid on Day 8, followed by five subsequent 100 mg gluteal injections every 28 days. The primary objective was to demonstrate steady-state bioequivalence. The primary endpoints were key pharmacokinetic parameters of paliperidone, including steady-state maximum concentration (Cmax,ss) and the area under the concentration-time curve over a dosing interval at steady state (AUCτ,ss). Bioequivalence was shown if the 90% confidence interval (CI) for the ratio of the geometric least squares means of the pharmacokinetic parameters (AUCτ,ss and Cmax,ss) fell within 80%-125%.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years inclusive at the time of consent.
2. Diagnosis of schizophrenia (ICD-10 criteria) prior to screening.
3. PANSS total score ≤70 at screening and at baseline.
4. CGI-S score ≤4 at screening and at baseline.
5. Body weight at screening: ≥50.0 kg (male) or ≥45.0 kg (female); body mass index (BMI) 19.0 to 35.0 kg/m2 (inclusive).
6. The participant and/or partner have no plans for pregnancy during the study and for 6 months after the last dose, and agree to use effective contraception (oral contraceptives are not allowed).
7. Signed informed consent and willingness and ability to comply with all study requirements.

Exclusion Criteria:

1. Known or suspected hypersensitivity to the study drug (paliperidone palmitate) or any of its components.
2. Diagnosis per ICD-10 or DSM-5 of any psychiatric disorder other than schizophrenia.
3. Clinically significant diseases or abnormalities, as judged by the investigator, in the respiratory, cardiovascular, gastrointestinal, genitourinary, reproductive, nervous, endocrine, or immune systems that may affect participant safety or interfere with study participation.
4. Laboratory abnormalities at screening or baseline meeting any of the following: (1) total bilirubin >1.5 × ULN, or AST or ALT >2 × ULN; (2) creatinine clearance (CLcr) <90 mL/min; (3) white blood cell count <3 × 10^9/L, or absolute neutrophil count <1.5 × 10^9/L, or platelets <80 × 10^9/L.
5. History of orthostatic hypotension or syncope due to orthostatic hypotension (except if stable for >6 months); or at screening/baseline, a decrease in systolic blood pressure ≥20 mmHg or diastolic blood pressure ≥10 mmHg within 3 minutes after changing from supine to standing.
6. Congenital long QT syndrome; uncontrolled or significant cardiovascular disease, including congestive heart failure of NYHA class II or higher, unstable angina, or myocardial infarction within 6 months prior to first study dose; significant arrhythmias (including frequent premature ventricular contractions), or clinically significant arrhythmias requiring treatment at screening; QTc >450 ms (male) or >460 ms (female) at screening or baseline; risk factors for torsades de pointes or sudden death (e.g., bradycardia, clinically significant hypokalemia or hypomagnesemia, current use of medications that prolong QTc); or other clinically significant ECG abnormalities as judged by the investigator.
7. Past or current neuroleptic malignant syndrome.
8. Parkinson's disease, Lewy body dementia, or dementia-related psychosis.
9. Past or current seizure or convulsive disorders (except childhood febrile seizures), or stroke or transient ischemic attack within 1 year prior to consent.
10. History of tardive dyskinesia induced by risperidone, paliperidone, or other antipsychotics.
11. Uncontrolled diabetes mellitus, or HbA1c ≥7% at screening or baseline.
12. Electroconvulsive therapy within 28 days prior to consent.
13. Blood loss ≥400 mL within 3 months prior to consent, or ≥200 mL within 1 month prior to consent due to donation, surgery, or other causes.
14. Esophageal motility disorders, dysphagia, or other conditions that confer risk of aspiration pneumonia.
15. Positive tests for hepatitis B surface antigen, hepatitis C antibody, HIV antibody, or treponemal (syphilis) antibody.
16. Harmful alcohol use: >14 units per week (1 unit = 360 mL beer, or 150 mL wine, or 45 mL spirits).
17. Use of any investigational drug within 1 month prior to first study dose (excluding paliperidone palmitate or placebo), or prior participation in a gene therapy or cell therapy clinical trial such that, in the investigator's judgment, the participant is not suitable for this study.
18. Major surgery within 3 months prior to consent, or planned surgery within 1 month after study completion.
19. High suicide risk: C-SSRS suicidal ideation items 4 or 5 answered "Yes" within the past 6 months at screening/baseline; or suicidal behavior within the past 6 months; or, in the investigator's judgment, a serious risk of suicide.
20. Prohibited medications/treatments: (1) ziprasidone or thioridazine within 4 weeks prior to consent; (2) any other long-acting injectable antipsychotic received within one labeled dosing interval prior to consent (except risperidone microspheres), or receipt of risperidone microspheres (e.g., Hengde®) within 6 weeks prior to consent; (3) non-selective or irreversible monoamine oxidase inhibitors within 1 month prior to first dose; (4) strong or moderate inhibitors or inducers of CYP3A4, CYP2D6, or P-gp within 2 weeks prior to consent.
21. Pregnant, breastfeeding, or planning pregnancy; except for women who are postmenopausal for ≥1 year or surgically sterile (e.g., bilateral tubal ligation with non-recanalized tubes, bilateral oophorectomy, or hysterectomy).
22. Drug abuse history, illicit drug use, or positive drug abuse screening within 1 year prior to consent.
23. Clinically significant history of syncope related to needles or blood draws. Any other condition that, in the investigator's opinion, makes the participant unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Title:Steady-State Peak Concentration (Cmax,ss) of Paliperidone After Intramuscular Administration. | Day148~Day176
  Steady-state maximum plasma concentration (Cmax,ss) will be determined to assess bioequivalence between the test and reference formulations of paliperidone palmitate injection after multiple intramuscular doses in patients with schizophrenia.
Area Under the Concentration-Time Curve over Dosing Interval (AUCτ,ss) of Paliperidone After Intramuscular Administration. | Day148~Day176
  Area under the plasma concentration-time curve during the dosing interval (AUCτ,ss) will be determined to assess bioequivalence between the test and reference formulations of paliperidone palmitate injection after multiple intramuscular doses in patients with schizophrenia.

SECONDARY OUTCOMES:
Steady-State Trough Concentration (Ctau,ss) | Day1~Day176
  Steady-state plasma trough concentration (Ctau,ss) of paliperidone will be measured to further characterize pharmacokinetics and assess bioequivalence between test and reference group.
Steady-State Average Concentration (Cav,ss) | Day1~Day176
  Average plasma concentration during the dosing interval (Cav,ss) will be evaluated at steady state.
Steady-State Minimum Concentration (Cmin,ss) | Day1~Day176
  Minimum plasma concentration during the dosing interval (Cmin,ss) at steady state will be determined.
Time to Maximum Concentration at Steady State (Tmax,ss) | Day1~Day176
  The time to reach maximum plasma concentration (Tmax,ss) will be assessed at steady state.
Degree of Fluctuation (DF) and Swing at Steady State | Day1~Day176
  The degree of fluctuation (DF) and swing of paliperidone plasma concentrations will be calculated at steady state.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Day1~Day176
  Number and percentage of participants experiencing ≥1 treatment-emergent adverse event (TEAE) after first dose; events coded by MedDRA (System Organ Class and Preferred Term); severity (mild/moderate/severe) and relationship to study drug assessed by investigator.
Number of Participants With Serious Adverse Events (SAEs) | Day1~Day176
  Number and percentage of participants experiencing ≥1 SAE, defined per ICH-GCP criteria; events coded by MedDRA (SOC/PT).
Clinical Global Impression-Severity (CGI-S) | Day1~Day176
  Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score Mean (SD) change in CGI-S score from baseline to end of treatment. Clinical Global Impression - Severity (CGI-S): The Clinical Global Impression - Severity Scale ranges from 1 to 7 (1 = normal, not at all ill; 7 = among the most extremely ill), and higher scores indicate worse clinical severity (worse outcome).
Proportion of Participants With Suicidal Ideation or Behavior (C-SSRS) | Day1~Day176
  Number and percentage of participants with suicidal ideation (items 4 or 5) and/or any suicidal behavior on the Columbia-Suicide Severity Rating Scale (C-SSRS).
  Columbia-Suicide Severity Rating Scale (C-SSRS): The Columbia-Suicide Severity Rating Scale rates suicidal ideation severity from 1 to 5 (0 = no suicidal ideation; 5 = most severe ideation), while suicidal behavior is recorded as present/absent; higher ideation category indicates a worse outcome (greater suicide risk).
Change From Baseline in Barnes Akathisia Rating Scale (BARS) Global Score | Day1~Day176
  Mean (SD) change in BARS global score from baseline to end of treatment. Barnes Akathisia Rating Scale (BARS): The Barnes Akathisia Rating Scale global score ranges from 0 to 5 (0 = no akathisia; 5 = severe akathisia), and higher scores indicate more severe akathisia (worse outcome).
Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score | Day1~Day176
  Mean (SD) change in AIMS total score from baseline to end of treatment. Abnormal Involuntary Movement Scale (AIMS): The Abnormal Involuntary Movement Scale total score commonly uses the sum of items 1-7 and ranges from 0 to 28 (0 = no abnormal movements; 28 = maximum severity on rated items); higher scores indicate more severe abnormal involuntary movements (worse outcome).
Change From Baseline in Simpson-Angus Scale (SAS) Total Score | Day1~Day176
  Mean (SD) change in SAS total score from baseline to end of treatment. Simpson-Angus Scale (SAS): The Simpson-Angus Scale total score ranges from 0 to 40 (10 items each scored 0-4), and higher scores indicate more severe drug-induced parkinsonism (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, M.D., Study Chair — Beijing Anding Hospital Capital Medical University
Locations (1):
- Beijing Anding Hospital Capital Medical University, Beijing, Beijing Municipality, China